CLINICAL TRIAL: NCT04690088
Title: Remifentanilio Titravimo būdų Palyginimas, Remiantis pacientų Budimo Kokybe Ligotai Nutukusiems Pacientams po laparoskopinių skrandžio tūrio mažinimo operacijų
Brief Title: Remifentanil Dosing Regimes for Anesthesia in Bariatric Surgery: Characteristics of Early Recovery
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Paulina Aldakauskaite, resident doctor, Lithuanian University of Health Sciences
Other Study IDs: BEC - MF - 93
Record Dates: First submitted 2020-10-08; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; remifentanil; manual infusion; target - controlled infusion
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manual infusion (control) group
- TCI (case) group

SUMMARY:
Early recovery characteristics are important for patients' safety and operating room turnover. Our aim was to compare fundamental methods for dosing remifentanil during morbid obesity surgeries: a manual infusion and a target-controlled infusion (TCI). Throughout study, patient's recovery time was tracked and compared between the groups.

DETAILED DESCRIPTION:
Introduction: The population of overweighted patients is increasing dramatically, therefore physicians face them in their daily practice (1-2). There are many guidelines showing the dose counting methods of intravenous anesthetics, but none of them are perfectly good for morbidity obese patients (3). Early recovery characteristics are important for patients' safety and operating room turnover (4).

Aim: Our aim was to compare fundamental methods for dosing remifentanil during morbid obesity surgeries: a manual infusion and a target-controlled infusion (TCI). Throughout study, patient's recovery time was tracked and compared between the groups.

Methods: 31 patients were evaluated who underwent bariatric surgery in Hospital of Lithuanian University of Health Sciences. All of them had received sevoflurane/remifentanil anaesthesia. Remifentanil infusion was randomly assigned to a manual (control group) or to a TCI (case group) method. We had evaluated patients' hemodynamics (arterial blood pressure, heart rate, saturation), spontaneous breathing and airway reflexes recovery time, time of extubation, eye opening, recovery of orientation and start of the following oral command. Also we had registered concentrations of remifentanil in the blood (according to automatic infusion pump) while using TCI method.

ELIGIBILITY:
Inclusion Criteria:

* Morbid patients to whom, according guidelines (BMI > 45 or BMI > 35 and chronic disease) bariatric surgery is indicated.
* Patient's approval.

Exclusion Criteria:

* Patients, younger than 18 years old.
* Patients who are higher than III ASA class.
* Patients who have higher sensibility to medications that are used during anesthesia.
* Patients with phycological disorders.
* Patients who can not fully communicate because of language barriers.
* Patients with surgical complications.
* Patient's disapproval.

Ages: 28 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with morbid obesity who are hospitalised in Hospital of Lithuanian University of Health Sciences Kaunas Clinics for laparoscopic bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
eye opening | up to 20 minutes
  The time of patient's respond after the end of remifentanyl infusion
spontaneous breathing | up to 20 minutes
  The time of patient's respond after the end of remifentanyl infusion
airway reflexes | up to 20 minutes
  The time of patient's respond after the end of remifentanyl infusion
orientation | up to 20 minutes
  The time of patient's respond after the end of remifentanyl infusion
oral command | 2,4,6,8,10,12,14,16,18,20 minutes
  The time of patient's respond after the end of remifentanyl infusion

SECONDARY OUTCOMES:
Heart rate | up to 20 minutes
  Measure was started after the end of remifentanyl infusion
Arterial blood pressure | up to 20 minutes
  Measure was started after the end of remifentanyl infusion
Saturation | up to 20 minutes
  Measure was started to record after the end of remifentanyl infusion
Remifentanyl dose | up to 20 minutes after surgery
  The amount of medication used during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clinical Guidelines on the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults--The Evidence Report. National Institutes of Health. Obes Res. 1998 Sep;6 Suppl 2:51S-209S. No abstract available. PMID 9813653
- [Background] Cheymol G. Effects of obesity on pharmacokinetics implications for drug therapy. Clin Pharmacokinet. 2000 Sep;39(3):215-31. doi: 10.2165/00003088-200039030-00004. PMID 11020136
- [Background] Adams JP, Murphy PG. Obesity in anaesthesia and intensive care. Br J Anaesth. 2000 Jul;85(1):91-108. doi: 10.1093/bja/85.1.91. No abstract available. PMID 10927998
- [Background] Michelsen LG, Hug CC Jr. The pharmacokinetics of remifentanil. J Clin Anesth. 1996 Dec;8(8):679-82. doi: 10.1016/s0952-8180(96)00179-1. PMID 8982900
- [Background] Egan TD, Kern SE, Muir KT, White J. Remifentanil by bolus injection: a safety, pharmacokinetic, pharmacodynamic, and age effect investigation in human volunteers. Br J Anaesth. 2004 Mar;92(3):335-43. doi: 10.1093/bja/aeh075. PMID 14970134
- See also: Cortrnez L I, Anderson B J. Current Opinion in Anaesthesiology 2018; 31(4):415-422. — https://www.ovid.com/product-details.496.html
- See also: Egan T D. Remyfentanil Pharmacocinetics and Pharmacodynamics. Clin. Pharmacokinet 1995; 29:80. — https://link.springer.com/article/10.2165/00003088-199529020-00003
- See also: Valstybinė vaistų kontrolės tarnyba. Remifentanil Kabi. — https://vapris.vvkt.lt/vvkt-web/public/medications/view/20375